CLINICAL TRIAL: NCT02542371
Title: Use of 99mTc Tilmanocept for Imaging Arterial Inflammation
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Navidea Biopharmaceuticals (Industry); Havard University Center for AIDS Research (Unknown)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2014P001832
Record Dates: First submitted 2015-08-26; First posted 2015-09-07 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: HIV
Keywords: HIV; Atherosclerosis; Tilmanocept
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, plasma and serum

GROUPS / COHORTS (4):
- HIV infected with known subclinical atherosclerosis
  Interventions: Other: Arterial Imaging
- HIV infected without known subclinical atherosclerosis
  Interventions: Other: Arterial Imaging
- Non-HIV infected with known subclinical atherosclerosis
  Interventions: Other: Arterial Imaging
- Non-HIV infected without known subclinical atherosclerosis
  Interventions: Other: Arterial Imaging

INTERVENTIONS:
Other: Arterial Imaging

SUMMARY:
The purpose of this study is to measure arterial 99mTc-Tilmanocept uptake using single photon emission computed tomography (SPECT/CT) scanning in HIV infected subjects known to have subclinical coronary atherosclerosis as assessed by contrast-enhanced coronary computed tomography angiography (CCTA).

DETAILED DESCRIPTION:
Detailed Description:

Patients with HIV have been shown to have increased atherosclerotic risk compared to age-matched controls, and this risk is thought to be related to increased systemic immune activation. Specifically, systemic immune activation may contribute to destabilizing coronary atherosclerotic plaque, leading to plaque rupture and myocardial infarction. This study is intended to measure arterial uptake of the macrophage specific marker 99mTc-Tilmanocept using single photon emission computed tomography, applied initially to a group of HIV-infected patients with known subclinical coronary atherosclerosis on CCTA. Moreover, traditional markers of CVD risk and inflammatory markers will be assessed in relation to CV imaging outcomes. Positive findings in the index HIV group with known subclinical atherosclerosis will prompt subsequent study of three comparison groups, as above.

ELIGIBILITY:
HIV infected subjects with known subclinical atherosclerosis:

Inclusion criteria:

* men and women, ages 18+, with documented HIV infection
* current use of antiretroviral therapy (ART), with no changes to regimen within last 3 months
* history of subclinical atherosclerosis on CCTA

Exclusion criteria:

* pregnancy or breastfeeding
* known active opportunistic infection requiring ongoing medical therapy (not including Hepatitis B/C)
* CD4 count < 50 cells/mm3
* history of angina, myocardial infarction, acute coronary syndrome, or coronary artery stenting or surgery
* recent and/or current treatment with prescription, systemic steroids or anti-inflammatory/immune suppressant medical therapies
* current use of statin or use of statin for > 1 month within the last 6 months
* known allergy to dextrans and/or DPTA and/or radiometals and/or iodinated contrast media
* eGFR < 60 ml/min/1.73 m2 calculated by CDK-EPI
* contraindications to beta blockers or nitroglycerin
* significant radiation exposure (>2 CT angiograms) received within the past 12 months
* BMI > 35 kg/m2 or waist circumference > 70 cm (scanner limitations)

HIV infected subjects without known subclinical atherosclerosis:

Inclusion criteria:

* men and women, ages 18+, with documented HIV infection
* current use of antiretroviral therapy (ART), with no changes to regimen within last 3 months
* history of clean aorta/ coronaries on CCTA

Exclusion criteria:

- Same as exclusion criteria for HIV infected subjects with known subclinical atherosclerosis

HIV negative subjects with known subclinical atherosclerosis:

Inclusion criteria:

* men and women, ages 18+, without documented HIV infection
* history of subclinical atherosclerosis on CCTA

Exclusion criteria:

* pregnancy or breastfeeding
* history of angina, myocardial infarction, acute coronary syndrome, or coronary artery stenting or surgery
* recent and/or current treatment with prescription, systemic steroids or anti-inflammatory/immune suppressant medical therapies
* current use of statin or use of statin for > 1 month within the last 6 months
* known allergy to dextrans and/or DPTA and/or radiometals and/or iodinated contrast media
* eGFR < 60 ml/min/1.73 m2 calculated by CDK-EPI
* contraindications to beta blockers or nitroglycerin
* significant radiation exposure (>2 CT angiograms) received within the past 12 months
* BMI > 35 kg/m2 or waist circumference > 70 cm (scanner limitations)

HIV negative subjects without known subclinical atherosclerosis:

Inclusion criteria:

* men and women, ages 18+, without documented HIV infection
* history of clean aorta/coronaries on CCTA

Exclusion criteria:

- Same as exclusion criteria for HIV negative subjects with known subclinical atherosclerosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected subjects and HIV non-infected subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Aortic 99mTc-Tilmanocept uptake on SPECT/CT scanning in HIV Patients | within 6 weeks of screening visit

SECONDARY OUTCOMES:
Aortic plaque burden and morphology on CCTA in HIV Patients | within 6 weeks of screening visit
Traditional markers of cardiovascular disease (CVD) risk and inflammatory markers in relation to cardiovascular imaging outcomes | within 6 weeks of screening visit
Imaging assessments in the coronary vasculature in HIV patients | within 6 weeks of screening visit
Comparison of imaging assessments b/ HIV patients w/ known subclinical atherosclerosis, HIV patients w/o known subclinical atherosclerosis, non HIV patients w/ known subclinical atherosclerosis and non HIV patients w/o known subclinical atherosclerosis | within 6 weeks of screening visit
99mTc-Tilmanocept uptake on SPECT/CT in regions other than the aorta | within 6 weeks of screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Toribio M, Wilks MQ, Hedgire S, Lu MT, Cetlin M, Wang M, Alhallak I, Durbin CG, White KS, Wallis Z, Schnittman SR, Stanley TL, El-Fakhri G, Lee H, Autissier P, Zanni MV, Williams KC, Grinspoon SK. Increased Macrophage-Specific Arterial Infiltration Relates to Noncalcified Plaque and Systemic Immune Activation in People With Human Immunodeficiency Virus. J Infect Dis. 2022 Nov 11;226(10):1823-1833. doi: 10.1093/infdis/jiac301. PMID 35856671
- [Derived] Zanni MV, Toribio M, Wilks MQ, Lu MT, Burdo TH, Walker J, Autissier P, Foldyna B, Stone L, Martin A, Cope F, Abbruzzese B, Brady T, Hoffmann U, Williams KC, El-Fakhri G, Grinspoon SK. Application of a Novel CD206+ Macrophage-Specific Arterial Imaging Strategy in HIV-Infected Individuals. J Infect Dis. 2017 Apr 15;215(8):1264-1269. doi: 10.1093/infdis/jix095. PMID 28204544